CLINICAL TRIAL: NCT02295475
Title: Apixaban for the Secondary Prevention of Thromboembolism: a Prospective Randomized Outcome Pilot Study Among Patients With the AntiphosPholipid Syndrome
Brief Title: Apixaban for Secondary Prevention of Thromboembolism Among Patients With AntiphosPholipid Syndrome
Acronym: ASTRO-APS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Scott C. Woller, MD (Other)
Collaborators: Bristol-Myers Squibb (Industry); University of Utah (Other)
Responsible Party: Sponsor-Investigator, Scott C. Woller, MD, Co-Director Thrombosis Program, Intermountain Health Care, Inc.
Organization: Intermountain Health Care, Inc. (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CV185-357; 1040354 (Other: Intermountain Healthcare IRB)
Record Dates: First submitted 2014-11-18; First posted 2014-11-20 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Antiphospholipid Syndrome; Thrombosis
Keywords: Apixaban; Eliquis
MeSH Terms: conditions — Antiphospholipid Syndrome; Thrombosis | interventions — apixaban; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Apixaban (Experimental): Subjects will receive apixaban 5 mg tablets taken twice daily for the duration of the study.
  Interventions: Drug: Apixaban
- Warfarin (Active Comparator): Subjects will receive warfarin for the duration of the study, with the dose and frequency adjusted per clinician discretion to achieve an INR (International Normalized Ratio) between 2 and 4.
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Apixaban
  Other Names: Eliquis
  Arms: Apixaban
Drug: Warfarin
  Other Names: Coumadin
  Arms: Warfarin

SUMMARY:
This study is designed to compare the safety and effectiveness of two blood thinners, apixaban and warfarin, for the prevention of blood clots in patients who have a higher risk of blood clots than the general population, a condition called "antiphospholipid syndrome".

DETAILED DESCRIPTION:
This study is a prospective, open-label, blinded event, pilot study that will randomize patients with a history of venous thrombosis and antiphospholipid syndrome (APS) already receiving anticoagulation to either warfarin or apixaban. The study will assess the safety and efficacy of apixaban compared with adjusted dose warfarin for the prevention of recurrent thrombosis (defined as the aggregate of arterial or venous thrombosis) and vascular death. The primary efficacy outcome will be confirmed upon adjudication by a panel blinded to the treatment arm. The primary safety outcome will be major bleeding and clinically relevant non-major bleeding events. Patients who consent to study participation will be randomized to anticoagulation with adjusted dose warfarin sodium or apixaban 5 mg by mouth twice daily. This pilot study will also provide information and experience identifying, recruiting, enrolling and randomizing patients with APS and a history of venous thrombosis to anticoagulation with apixaban or warfarin for the prevention of recurrent thrombosis.

ELIGIBILITY:
Inclusion Criteria:

1. Be ≥ 18 years of age
2. Have a clinical diagnosis of the antiphospholipid syndrome (APS) and a history of venous thrombosis only (excluding arterial thrombosis as recommended by the Data Safety Monitoring Board (DSMB)) for which the patient is receiving anticoagulation therapy for the prevention of recurrent thrombosis;

   1. Anticoagulation is defined as warfarin sodium titrated at the discretion of the clinician to a target INR (International Normalized Ratio) 2.5 (range 2-3), 3.0 (range 2.5-3.5), or 3.5 (range 3-4).
   2. Should the patient be receiving some other form of anticoagulation (apixaban, rivaroxaban, edoxaban, dabigatran etexilate, low-molecular weight heparin) and is willing to be randomized to warfarin with a target INR 2.5 or apixaban 5 mg by mouth twice daily and meets all other inclusion criteria.
3. Able to undergo magnetic resonance imaging (MRI) of the brain;
4. Have completed at least 6 months of anticoagulation for the indication of venous thrombosis and be without symptoms or signs consistent with acute thrombosis for a minimum of 6 months;
5. Be willing to provide informed consent to contact the subjects anticoagulation provider for INRs and dosing as well as details regarding any adverse events;
6. A woman of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of hCG (Human Chorionic Gonadotropin) within 24 hours prior to the start of study drug;
7. Women must not be breastfeeding;
8. A WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug apixaban plus 5 half-lives of study drug apixaban (3 days) plus 30 days (duration of ovulatory cycle) for a total of 33 days post-treatment completion;
9. Males who are sexually active with any WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug apixaban plus 5 half-lives of the study drug apixaban (3 days) plus 90 days (duration of sperm turnover) for a total of 93 days post-treatment completion;
10. Azoospermic males and women who are continuously not heterosexually active are exempt from contraceptive requirements. However, a WOCBP must still undergo pregnancy testing as described above;
11. If they are actively receiving a strong dual inhibitor of cytochrome P450 3A4 (CYP3A4) and P-gp, such as ketoconazole, itraconazole, ritonavir, and are agreeable to taking apixaban 2.5 mg twice daily.

Exclusion Criteria:

1. A history of arterial thromboembolism (e.g., stroke, myocardial infarction, or other arterial thrombosis);
2. Another indication for long-term anticoagulation for which no FDA (Food & Drug Administration) approval of apixaban exists (e.g., mechanical heart valve);
3. A life expectancy of less than 1 year;
4. Is unable to attend follow-up appointments;
5. Is participating in a clinical trial or has participated in a trial within the last 30 days;
6. Is receiving concomitant dual antiplatelet therapy;
7. Requires aspirin dose of greater than 165 mg daily;
8. Requires clopidogrel, ticagrelor, prasugrel, or another P2Y12 inhibitor;
9. A hemoglobin level of less than 8 mg per deciliter;
10. A platelet count of less than 50,000 per cubic millimeter;
11. Serum creatinine level of more than 2.5 mg per deciliter or a calculated creatinine clearance of less than 25 ml per minute;
12. Alanine aminotransferase or aspartate aminotransferase level greater than 2 times the upper limit of the normal range;
13. A total bilirubin more than 1.5 times the upper limit of the normal range;
14. Have active cancer for which treatment (chemotherapy/radiation therapy) is being delivered or has been delivered within the last 3 months;
15. Are actively taking a strong dual inducer of CYP3A4 and P-gp, such as:

    * rifampin
    * carbamazepine
    * phenytoin
    * St.John's wort
16. Intend pregnancy or breastfeeding within the next year;
17. Have a known allergy to apixaban, rivaroxaban, or edoxaban;
18. Have experienced thrombosis while receiving warfarin at a target INR of 2 to 3 and have been assigned a higher target INR at the discretion of the treating clinician;
19. Have active pathological bleeding;
20. Have a history of catastrophic APS (CAPS) as defined by clinical routine;
21. At the discretion of the investigator, are not considered to be good candidates secondary to a safety concern.

Patients who meet the above inclusion & exclusion criteria will be offered participation in the study. After informed consent is obtained, the patient will be consented for Magnetic Resonance Imaging (MRI). A brain MRI without contrast including weighted imaging and fluid-attenuated inversion recovery (FLAIR) will be performed as a study procedure to rule out prior stroke. If the patient has radiographic evidence of prior stroke on this MRI, then the patient will not be randomized, and will not be included in future study procedures or study analyses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-12-10 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
Rate (number divided by duration) of clinically overt thromboses (arterial and/or venous) or vascular death | From time of first dose of study drug through 2 days after receiving the last dose of study drug at the end of 12 months of treatment
Rate (number divided by duration) of occurrence of major (including fatal) and clinically relevant non-major bleeding | From time of first dose of study drug through 2 days after receiving the last dose of study drug at the end of 12 months of treatment
  Major bleeding is clinically overt bleeding accompanied by one or more of the following: a decrease in the hemoglobin level of 2 g per deciliter or more, transfusion of 2 or more units of packed red cells, bleeding at a critical site (intracranial, intraspinal, intraocular, pericardial, intraarticular, intramuscular with compartment syndrome, or retroperitoneal), or fatal bleeding. Clinically relevant non-major bleeding is defined as clinically overt bleeding that does not satisfy the criteria for major bleeding and that led to hospital admission, physician-guided medical or surgical treatment, or a change in antithrombotic therapy.

SECONDARY OUTCOMES:
Net clinical benefit (combination of occurrence of thrombosis and bleeding rates) | From time of first dose of study drug through 2 days after receiving the last dose of study drug at the end of 12 months of treatment
  Sum of number of thrombosis and bleeding events divided by duration

CONTACTS AND LOCATIONS:
Overall Officials: Scott C Woller, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (2):
- United States (2):
  - The James Comprehensive Cancer Center, Columbus, Ohio
  - Intermountain Medical Center, Murray, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miyakis S, Lockshin MD, Atsumi T, Branch DW, Brey RL, Cervera R, Derksen RH, DE Groot PG, Koike T, Meroni PL, Reber G, Shoenfeld Y, Tincani A, Vlachoyiannopoulos PG, Krilis SA. International consensus statement on an update of the classification criteria for definite antiphospholipid syndrome (APS). J Thromb Haemost. 2006 Feb;4(2):295-306. doi: 10.1111/j.1538-7836.2006.01753.x. PMID 16420554
- [Background] Agnelli G, Buller HR, Cohen A, Curto M, Gallus AS, Johnson M, Porcari A, Raskob GE, Weitz JI; AMPLIFY-EXT Investigators. Apixaban for extended treatment of venous thromboembolism. N Engl J Med. 2013 Feb 21;368(8):699-708. doi: 10.1056/NEJMoa1207541. Epub 2012 Dec 8. PMID 23216615
- [Background] Agnelli G, Buller HR, Cohen A, Curto M, Gallus AS, Johnson M, Masiukiewicz U, Pak R, Thompson J, Raskob GE, Weitz JI; AMPLIFY Investigators. Oral apixaban for the treatment of acute venous thromboembolism. N Engl J Med. 2013 Aug 29;369(9):799-808. doi: 10.1056/NEJMoa1302507. Epub 2013 Jul 1. PMID 23808982
- [Background] Connolly SJ, Eikelboom J, Joyner C, Diener HC, Hart R, Golitsyn S, Flaker G, Avezum A, Hohnloser SH, Diaz R, Talajic M, Zhu J, Pais P, Budaj A, Parkhomenko A, Jansky P, Commerford P, Tan RS, Sim KH, Lewis BS, Van Mieghem W, Lip GY, Kim JH, Lanas-Zanetti F, Gonzalez-Hermosillo A, Dans AL, Munawar M, O'Donnell M, Lawrence J, Lewis G, Afzal R, Yusuf S; AVERROES Steering Committee and Investigators. Apixaban in patients with atrial fibrillation. N Engl J Med. 2011 Mar 3;364(9):806-17. doi: 10.1056/NEJMoa1007432. Epub 2011 Feb 10. PMID 21309657
- [Background] Granger CB, Alexander JH, McMurray JJ, Lopes RD, Hylek EM, Hanna M, Al-Khalidi HR, Ansell J, Atar D, Avezum A, Bahit MC, Diaz R, Easton JD, Ezekowitz JA, Flaker G, Garcia D, Geraldes M, Gersh BJ, Golitsyn S, Goto S, Hermosillo AG, Hohnloser SH, Horowitz J, Mohan P, Jansky P, Lewis BS, Lopez-Sendon JL, Pais P, Parkhomenko A, Verheugt FW, Zhu J, Wallentin L; ARISTOTLE Committees and Investigators. Apixaban versus warfarin in patients with atrial fibrillation. N Engl J Med. 2011 Sep 15;365(11):981-92. doi: 10.1056/NEJMoa1107039. Epub 2011 Aug 27. PMID 21870978
- [Background] Cano SJ, Lamping DL, Bamber L, Smith S. The Anti-Clot Treatment Scale (ACTS) in clinical trials: cross-cultural validation in venous thromboembolism patients. Health Qual Life Outcomes. 2012 Sep 26;10:120. doi: 10.1186/1477-7525-10-120. PMID 23013426
- [Background] Bamber L, Wang MY, Prins MH, Ciniglio C, Bauersachs R, Lensing AW, Cano SJ. Patient-reported treatment satisfaction with oral rivaroxaban versus standard therapy in the treatment of acute symptomatic deep-vein thrombosis. Thromb Haemost. 2013 Oct;110(4):732-41. doi: 10.1160/TH13-03-0243. Epub 2013 Jul 11. PMID 23846019
- [Background] Cohen H, Machin SJ. Antithrombotic treatment failures in antiphospholipid syndrome: the new anticoagulants? Lupus. 2010 Apr;19(4):486-91. doi: 10.1177/0961203310361355. PMID 20353992
- [Background] Alarcon-Segovia D, Perez-Vazquez ME, Villa AR, Drenkard C, Cabiedes J. Preliminary classification criteria for the antiphospholipid syndrome within systemic lupus erythematosus. Semin Arthritis Rheum. 1992 Apr;21(5):275-86. doi: 10.1016/0049-0172(92)90021-5. PMID 1604324
- [Background] Asherson RA, Khamashta MA, Ordi-Ros J, Derksen RH, Machin SJ, Barquinero J, Outt HH, Harris EN, Vilardell-Torres M, Hughes GR. The "primary" antiphospholipid syndrome: major clinical and serological features. Medicine (Baltimore). 1989 Nov;68(6):366-74. PMID 2509856
- [Background] Vianna JL, Khamashta MA, Ordi-Ros J, Font J, Cervera R, Lopez-Soto A, Tolosa C, Franz J, Selva A, Ingelmo M, et al. Comparison of the primary and secondary antiphospholipid syndrome: a European Multicenter Study of 114 patients. Am J Med. 1994 Jan;96(1):3-9. doi: 10.1016/0002-9343(94)90108-2. PMID 8304360
- [Background] Cervera R, Serrano R, Pons-Estel GJ, Ceberio-Hualde L, Shoenfeld Y, de Ramon E, Buonaiuto V, Jacobsen S, Zeher MM, Tarr T, Tincani A, Taglietti M, Theodossiades G, Nomikou E, Galeazzi M, Bellisai F, Meroni PL, Derksen RH, de Groot PG, Baleva M, Mosca M, Bombardieri S, Houssiau F, Gris JC, Quere I, Hachulla E, Vasconcelos C, Fernandez-Nebro A, Haro M, Amoura Z, Miyara M, Tektonidou M, Espinosa G, Bertolaccini ML, Khamashta MA; Euro-Phospholipid Project Group (European Forum on Antiphospholipid Antibodies). Morbidity and mortality in the antiphospholipid syndrome during a 10-year period: a multicentre prospective study of 1000 patients. Ann Rheum Dis. 2015 Jun;74(6):1011-8. doi: 10.1136/annrheumdis-2013-204838. Epub 2014 Jan 24. PMID 24464962
- [Background] Galli M, Luciani D, Bertolini G, Barbui T. Anti-beta 2-glycoprotein I, antiprothrombin antibodies, and the risk of thrombosis in the antiphospholipid syndrome. Blood. 2003 Oct 15;102(8):2717-23. doi: 10.1182/blood-2002-11-3334. Epub 2003 Jun 19. No abstract available. PMID 12816875
- [Background] Rosamond W, Flegal K, Furie K, Go A, Greenlund K, Haase N, Hailpern SM, Ho M, Howard V, Kissela B, Kittner S, Lloyd-Jones D, McDermott M, Meigs J, Moy C, Nichol G, O'Donnell C, Roger V, Sorlie P, Steinberger J, Thom T, Wilson M, Hong Y; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2008 update: a report from the American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Circulation. 2008 Jan 29;117(4):e25-146. doi: 10.1161/CIRCULATIONAHA.107.187998. Epub 2007 Dec 17. No abstract available. PMID 18086926
- [Background] Crowther MA, Ginsberg JS, Julian J, Denburg J, Hirsh J, Douketis J, Laskin C, Fortin P, Anderson D, Kearon C, Clarke A, Geerts W, Forgie M, Green D, Costantini L, Yacura W, Wilson S, Gent M, Kovacs MJ. A comparison of two intensities of warfarin for the prevention of recurrent thrombosis in patients with the antiphospholipid antibody syndrome. N Engl J Med. 2003 Sep 18;349(12):1133-8. doi: 10.1056/NEJMoa035241. PMID 13679527
- [Background] Petri M. Thrombosis and systemic lupus erythematosus: the Hopkins Lupus Cohort perspective. Scand J Rheumatol. 1996;25(4):191-3. doi: 10.3109/03009749609069986. PMID 8792794
- [Background] Witt DM, Sadler MA, Shanahan RL, Mazzoli G, Tillman DJ. Effect of a centralized clinical pharmacy anticoagulation service on the outcomes of anticoagulation therapy. Chest. 2005 May;127(5):1515-22. doi: 10.1378/chest.127.5.1515. PMID 15888822
- [Background] van Walraven C, Jennings A, Oake N, Fergusson D, Forster AJ. Effect of study setting on anticoagulation control: a systematic review and metaregression. Chest. 2006 May;129(5):1155-66. doi: 10.1378/chest.129.5.1155. PMID 16685005
- [Background] Hansson L, Hedner T, Dahlof B. Prospective randomized open blinded end-point (PROBE) study. A novel design for intervention trials. Prospective Randomized Open Blinded End-Point. Blood Press. 1992 Aug;1(2):113-9. doi: 10.3109/08037059209077502. PMID 1366259
- [Background] Connolly SJ, Ezekowitz MD, Yusuf S, Eikelboom J, Oldgren J, Parekh A, Pogue J, Reilly PA, Themeles E, Varrone J, Wang S, Alings M, Xavier D, Zhu J, Diaz R, Lewis BS, Darius H, Diener HC, Joyner CD, Wallentin L; RE-LY Steering Committee and Investigators. Dabigatran versus warfarin in patients with atrial fibrillation. N Engl J Med. 2009 Sep 17;361(12):1139-51. doi: 10.1056/NEJMoa0905561. Epub 2009 Aug 30. PMID 19717844
- [Background] Cohen AT, Spiro TE, Buller HR, Haskell L, Hu D, Hull R, Mebazaa A, Merli G, Schellong S, Spyropoulos A, Tapson V. Extended-duration rivaroxaban thromboprophylaxis in acutely ill medical patients: MAGELLAN study protocol. J Thromb Thrombolysis. 2011 May;31(4):407-16. doi: 10.1007/s11239-011-0549-x. PMID 21359646
- [Background] EINSTEIN-PE Investigators; Buller HR, Prins MH, Lensin AW, Decousus H, Jacobson BF, Minar E, Chlumsky J, Verhamme P, Wells P, Agnelli G, Cohen A, Berkowitz SD, Bounameaux H, Davidson BL, Misselwitz F, Gallus AS, Raskob GE, Schellong S, Segers A. Oral rivaroxaban for the treatment of symptomatic pulmonary embolism. N Engl J Med. 2012 Apr 5;366(14):1287-97. doi: 10.1056/NEJMoa1113572. Epub 2012 Mar 26. PMID 22449293
- [Background] Lassen MR, Ageno W, Borris LC, Lieberman JR, Rosencher N, Bandel TJ, Misselwitz F, Turpie AG; RECORD3 Investigators. Rivaroxaban versus enoxaparin for thromboprophylaxis after total knee arthroplasty. N Engl J Med. 2008 Jun 26;358(26):2776-86. doi: 10.1056/NEJMoa076016. PMID 18579812
- [Background] Rosove MH, Brewer PM. Antiphospholipid thrombosis: clinical course after the first thrombotic event in 70 patients. Ann Intern Med. 1992 Aug 15;117(4):303-8. doi: 10.7326/0003-4819-117-4-303. PMID 1637025
- [Background] Khamashta MA, Cuadrado MJ, Mujic F, Taub NA, Hunt BJ, Hughes GR. The management of thrombosis in the antiphospholipid-antibody syndrome. N Engl J Med. 1995 Apr 13;332(15):993-7. doi: 10.1056/NEJM199504133321504. PMID 7885428
- [Background] Ruiz-Irastorza G, Khamashta MA, Hunt BJ, Escudero A, Cuadrado MJ, Hughes GR. Bleeding and recurrent thrombosis in definite antiphospholipid syndrome: analysis of a series of 66 patients treated with oral anticoagulation to a target international normalized ratio of 3.5. Arch Intern Med. 2002 May 27;162(10):1164-9. doi: 10.1001/archinte.162.10.1164. PMID 12020188
- [Background] Keeling D, Mackie I, Moore GW, Greer IA, Greaves M; British Committee for Standards in Haematology. Guidelines on the investigation and management of antiphospholipid syndrome. Br J Haematol. 2012 Apr;157(1):47-58. doi: 10.1111/j.1365-2141.2012.09037.x. Epub 2012 Feb 8. No abstract available. PMID 22313321
- [Background] Giannakopoulos B, Krilis SA. How I treat the antiphospholipid syndrome. Blood. 2009 Sep 3;114(10):2020-30. doi: 10.1182/blood-2009-05-220756. Epub 2009 Jul 8. PMID 19587374
- [Background] Les I, Ruiz-Irastorza G, Khamashta MA. Intensity and duration of anticoagulation therapy in antiphospholipid syndrome. Semin Thromb Hemost. 2012 Jun;38(4):339-47. doi: 10.1055/s-0032-1304720. Epub 2012 Mar 30. PMID 22467528
- [Background] Nayer A, Ortega LM. Catastrophic antiphospholipid syndrome: a clinical review. J Nephropathol. 2014 Jan;3(1):9-17. doi: 10.12860/jnp.2014.03. Epub 2014 Jan 1. PMID 24644537
- [Background] Rosendaal FR, Cannegieter SC, van der Meer FJ, Briet E. A method to determine the optimal intensity of oral anticoagulant therapy. Thromb Haemost. 1993 Mar 1;69(3):236-9. PMID 8470047
- [Background] Cronan JJ. Venous thromboembolic disease: the role of US. Radiology. 1993 Mar;186(3):619-30. doi: 10.1148/radiology.186.3.8430164.
- [Background] Prandoni P, Cogo A, Bernardi E, Villalta S, Polistena P, Simioni P, Noventa F, Benedetti L, Girolami A. A simple ultrasound approach for detection of recurrent proximal-vein thrombosis. Circulation. 1993 Oct;88(4 Pt 1):1730-5. doi: 10.1161/01.cir.88.4.1730. PMID 8403319
- [Background] Bates SM, Jaeschke R, Stevens SM, Goodacre S, Wells PS, Stevenson MD, Kearon C, Schunemann HJ, Crowther M, Pauker SG, Makdissi R, Guyatt GH. Diagnosis of DVT: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e351S-e418S. doi: 10.1378/chest.11-2299. PMID 22315267
- [Background] Stein PD, Gottschalk A, Sostman HD, Chenevert TL, Fowler SE, Goodman LR, Hales CA, Hull RD, Kanal E, Leeper KV Jr, Nadich DP, Sak DJ, Tapson VF, Wakefield TW, Weg JG, Woodard PK. Methods of Prospective Investigation of Pulmonary Embolism Diagnosis III (PIOPED III). Semin Nucl Med. 2008 Nov;38(6):462-70. doi: 10.1053/j.semnuclmed.2008.06.003. PMID 19331840
- [Background] PIOPED Investigators. Value of the ventilation/perfusion scan in acute pulmonary embolism. Results of the prospective investigation of pulmonary embolism diagnosis (PIOPED). JAMA. 1990 May 23-30;263(20):2753-9. doi: 10.1001/jama.1990.03440200057023. PMID 2332918
- [Background] van Belle A, Buller HR, Huisman MV, Huisman PM, Kaasjager K, Kamphuisen PW, Kramer MH, Kruip MJ, Kwakkel-van Erp JM, Leebeek FW, Nijkeuter M, Prins MH, Sohne M, Tick LW; Christopher Study Investigators. Effectiveness of managing suspected pulmonary embolism using an algorithm combining clinical probability, D-dimer testing, and computed tomography. JAMA. 2006 Jan 11;295(2):172-9. doi: 10.1001/jama.295.2.172. PMID 16403929
- [Background] Schulman S, Kearon C; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in non-surgical patients. J Thromb Haemost. 2005 Apr;3(4):692-4. doi: 10.1111/j.1538-7836.2005.01204.x. PMID 15842354
- [Derived] Woller SC, Stevens SM, Kaplan D, Wang TF, Branch DW, Groat D, Wilson EL, Armbruster B, Aston VT, Lloyd JF, Rondina MT, Elliott CG. Apixaban compared with warfarin to prevent thrombosis in thrombotic antiphospholipid syndrome: a randomized trial. Blood Adv. 2022 Mar 22;6(6):1661-1670. doi: 10.1182/bloodadvances.2021005808. PMID 34662890